CLINICAL TRIAL: NCT04996992
Title: Multimodal Magnetic Resonance Imaging Study for MRgFUS Pallidothalamic Tractotomy for Therapy-Resistant Parkinson's Disease
Brief Title: MRgFUS Pallidothalamic Tractotomy for Therapy-Resistant Parkinson's Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Xin Lou, Deputy Director of Department of Radiology, Chinese PLA General Hospital
Other Study IDs: MRgFUS-PTT-PD
Record Dates: First submitted 2021-07-31; First posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-07

CONDITIONS: Parkinson Disease; Magnetic Resonance Imaging
Keywords: MR-guided focused ultrasound; pallidothalamic tractotomy
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parkinson's disease: The cohort includes patients with Parkinson's disease who underwent MRgFUS pallidothalamic tractotomy (PTT).
  Interventions: Procedure: MR-guided focused ultrasound

INTERVENTIONS:
Procedure: MR-guided focused ultrasound — MR-guided focused ultrasound pallidothalamic tractotomy is a minimally invasive and effective procedure for thetreatment of Parkinson's disease(PD) patients.

SUMMARY:
To investigate the neural mechanism of Magnetic resonance-guided focused ultrasound (MRgFUS) Pallidothalamic Tractotomy in Parkinson's disease through multi-model MRI, and identify imaging biomarkers for triaging candidates and predicting the clinical outcomes.

Parkinson's disease (PD) is the second most progressive neurodegenerative disease with many motor and non-motor symptoms, which brings heavy burden to the family and the society.

MRgFUS pallidothalamic tractotomy allows to address all symptoms of PD without skull opening and with very limited tissue ablation, but with varying effectiveness. The unknown pathogenesis of PD has greatly contributed to this variance. Therefore, in order to optimize the clinical application of MRgFUS pallidothalamic tractotomy, it is important to reveal the pathogenesis of Parkinson's disease by using multiple modality MRI methods, and identify imaging biomarkers to triage suitable candidates and predict clinical outcomes.

DETAILED DESCRIPTION:
Treatment scheme:

All patients will first receive uni- or bilateral MRgFUS PTT. As to bilateral interventions, the second one will take place at least 6 months after the first PTT. Patients with unilateral intervention will be followed to 1 year. Patients with bilateral interventions will be followed to 1 year after the second intervention. Baseline clinical demographics, Unified Parkinson Disease Rating Scale (UPDRS), treatment parameters (energy, power, duration time, temperature, target location) , associated adverse effects were recorded.

Imaging protocols:

T2; T2 Flair; DWI; ESWAN; MRS; 3D ASL 2.0s; 3D-T1; DTI; rs-functional MRI

Imaging evaluation:

1. Lesion appearance and volume are measured by T2, T2 Flair, DWI, ESWAN, 3D-T1;
2. ESWAN and MRS manifests the changes of iron deposition and metabolism, respectively;
3. ASL shows regional cerebral blood flow associated with the procedure;
4. DTI demonstrates the destruction of white matter integrity.
5. Rs-functional MRI reflects alterations of resting-state brain activity.

Treatment:

MRgFUS pallidothalamic tractotomy

Follow-up:

MRI + clinical evaluation: Baseline, 3-day, 1-week, 1-month, 3-months, 6-months,12-months

ELIGIBILITY:
Inclusion Criteria:

1. Regardless of sex, aged 30 or above, hope to treat bilateral motor symptoms and receive the other side treatment plan at the 6th month;
2. Subjects are able and willing to give informed consent and can participate in whole study visits;
3. It was clinically diagnosed as Parkinson's disease and confirmed by functional neurosurgeons;
4. The subjects should respond to levodopa;
5. In the off-medication state, the subjects' MDS-UPDRS scores were 30 or more.

Exclusion Criteria:

1. The subjects scored 3 or more in the pull-back test;
2. Parkinson's disease symptoms were suspected as the side effects of antipsychotics;
3. severe cognitive impairment confirmed by neuropsychologists;
4. subjects with other neurodegenerative diseases;
5. Subjects with unstable mental illness, defined as active, uncontrolled depression, schizophrenia, delusions, hallucinations or suicide intention;
6. Pregnant or lactating women;
7. Subjects with alcohol or drug abuse;
8. Subjects with unstable heart condition or severe hypertension;
9. Subjects with a history of abnormal bleeding or clotting.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's disease
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2021-08-15 (Estimated); Primary Completion 2023-08-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
primary efficacy outcome | 1 year
  The primary endpoints at 6 months and 1 year postoperatively were the Unified Parkinson's Disease Rating Scale (UPDRS) scores.
primary safety outcome | 1 year
  Primary safety outcome was assessed by monitoring the incidence and severity of the procedure-related adverse events from the procedure through 1 year after treatment for all patients.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Lou, MD, Study Chair — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided